CLINICAL TRIAL: NCT03433040
Title: Impact of a Higher Dose on the Pharmacokinetics of 17-alpha Hydroxyprogesterone Caproate in Obese Women
Brief Title: 17OHP-C Dosing Among Obese Pregnant Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Anthony Odibo MD, Director Ultrasound and Fetal Therapy, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00026055
Record Dates: First submitted 2017-08-28; First posted 2018-02-14 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-11

CONDITIONS: Premature Birth; Absorption; Chemicals
MeSH Terms: conditions — Premature Birth | interventions — 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- non obese (Other): 250mg 17 OHP-C
  Interventions: Drug: 17-Hydroxyprogesterone Capronate
- obese - control (Other): 250mg 17 OHP-C
  Interventions: Drug: 17-Hydroxyprogesterone Capronate
- obese (Experimental): 500mg 17 OHP-C
  Interventions: Drug: 17-Hydroxyprogesterone Capronate

INTERVENTIONS:
Drug: 17-Hydroxyprogesterone Capronate — 17-Hydroxyprogesterone Capronate 250mg versus 500mg

SUMMARY:
Emergency data suggest 17OHP-C may be less efficacious in obese women. Since obesity is associated with lower levels of plasma 17OHP-C, the investigator hypothesize that higher doses of 17OHP-C may help to prevent spontaneous PTB among obese women. The study aims to compare the pharmacokinetics of 17 OHP-C in obese compared with non-obese women.

DETAILED DESCRIPTION:
Prospective three arm study of women with a prior spontaneous PTB. Non-obese women will receive the standard 250 mg weekly dose of 17 OHP-C while obese women will be randomly assigned to the standard (250 mg) or higher dose (500 mg). The resulting three groups will consist of:

1. Normal weight women on 250mg 17OHPC
2. Obese women on 250mg 17OHPC
3. Obese women on 500mg of 17OHPC

Initial Enrollment: Pregnant patients receiving prenatal care at one of the USF affiliated sites or Washington University in St. Louis sites who report a history of a PTB will be approached by the research nurse. The research nurse will explain the study, review inclusion/exclusion criteria with the patient, and invite interested potential study candidates to sign a medical records release so that records from the previous PTB can be reviewed. If the medical records confirm the birth of a previous PTB was of a live born singleton gestation between the gestational ages of 20 weeks and 36 weeks and 6 days then the patient will be invited to participate in the study. At that time the informed consent form will be thoroughly reviewed with the patient, and if the patient desires to enroll, the patient will provide informed consent to enroll in the study. Consecutive women with normal BMI or obese women meeting the inclusion criteria will be approached to avoid selection bias.

Randomization: will occur at the time of enrollment. The randomization will be computer generated. Randomization envelopes indicating the randomization arm will be prepared ahead of time and the next consecutive envelope will be used at time of enrollment.

Pharmacokinetic studies: Sampling schedule in order to investigate the pharmacokinetics of 250 mg 17OHP-C weekly as compared to 500 mg 17OHP-C weekly in obese women as well as 250 mg in non-obese women will be performed as follows:

- Using principles described by Caritis et al., four completed weeks of 17OHP-C therapy is required prior to sampling anticipating that steady state will be achieved by this time point.

ELIGIBILITY:
Inclusion Criteria:

* - Pregnant women, with a singleton gestation
* Ages 18 - 55
* Able to read and write in English and / or Spanish
* History of spontaneous PTB
* Obesity (≥ 30 kg / m2 ) vs non-obese groups (18 - 29.9 kg / m2 ) defined by first documented body mass index at an office visit
* Gestational age between 12 weeks, 0 days and 24 weeks, 6 days of gestation
* An ultrasound before 24 + 6 weeks gestation to confirm dating and to rule out major fetal anomalies
* Willing to have weekly injections at the physician's office
* The newborn will be enrolled on the mothers consent for chart review only

https://register.clinicaltrials.gov/prs/html/definitions.html?popup=true#Eligibility

Exclusion Criteria:

* - Multifetal gestation
* Known fetal anomaly
* Current progesterone treatment
* Known or suspected breast cancer, other hormone-sensitive cancer, or history of these conditions
* Current or history of thrombosis or thromboembolic disorder
* Current anticoagulation
* Undiagnosed abnormal vaginal bleeding unrelated to pregnancy
* Cholestatic jaundice of pregnancy
* Liver tumors, benign or malignant, or active liver disease
* uncontrolled hypertension (controlled hypertension is eligible)
* A seizure disorder
* Current or planned cervical cerclage
* Plan to deliver elsewhere

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony O Odibo, MD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - University of South Florida, Tampa, Florida
  - Washington University in St Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non Obese | Obese - Control | Obese
Started | 19 | 16 | 9
Completed | 17 | 8 | 5
Not Completed | 2 | 8 | 4

BASELINE CHARACTERISTICS:
Population: Study stopped due to futility with enrolling in the obese group with BMI > 30.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non Obese | Obese - Control | Obese | Total
Number analyzed (Participants) | 17 | 8 | 5 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 8 | 5 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (5.1) | 31.6 (6.4) | 31.4 (4.6) | 31.7 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 8 | 5 | 30
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 4 | 15
  White | 9 | 4 | 1 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants] — Number enrolled from different regions
  Participants
    United States | 17 | 8 | 5 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Trough Levels of 17-OHPC in the Three Groups at 20-22 Weeks, 27-29 Weeks and 34-36 Weeks.
Description: Blood levels
Time Frame: From enrollment to 36 weeks of pregnancy
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Non Obese | Obese - Control | Obese
Number analyzed (Participants) | 17 | 8 | 5
ng/ml
  20-22 weeks | 10.1 (4.5) | 13.0 (5.1) | 18.0 (6.7)
  27-29 weeks | 11.5 (4.8) | 8.1 (5.6) | 17.9 (2.5)
  34-36 weeks | 15.2 (12.5) | 11.1 (6.2) | 24.6 (7.1)

2. Secondary Outcome: Gestational Age at Delivery
Description: Gestational age at delivery in weeks . Too few to dichotomize to <37, 34 and 32 weeks as previously planned.
Time Frame: Up to 37 weeks
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Non Obese | Obese - Control | Obese
Number analyzed (Participants) | 17 | 8 | 5
Weeks | 36.7 (2.6) | 38.4 (1.4) | 32.2 (5.5)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Non Obese | Obese - Control | Obese
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/17 | 0/8 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT03433040/Prot_SAP_001.pdf